CLINICAL TRIAL: NCT07142967
Title: Trial Evaluating the Safety and Efficacy Of MR-Linac-Guided Radiotherapy as Salvage Treatment After External Beam Radiotherapy Recurrence (TUMORNATOR II)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-00856
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Intraprostatic Prostate Cancer
Keywords: prostate adenocarcinoma
MeSH Terms: interventions — Radiosurgery; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MRI-Linac-based SBRT with online adaptive replanning (Experimental): Participants will be treated with MR-guided stereotactic body radiation therapy/radiosurgery (SBRT) directed to the prostate using a 1.5 Tesla (1.5T) Elekta UNITY MR-Linac system in conjunction with 4-6 months of androgen deprivation therapy (ADT).
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT); Drug: Androgen Deprivation Therapy (ADT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — SBRT will be delivered with a prescription dose of 8 Gy x 5 fractions prescribed to the 95% isodose line encompassing the dominant recurrent intraprostatic lesion (DRIL) as seen on MRI and/or PET PSMA imaging plus 4mm (GTV+4mm=CTV_40). Remainder of the prostate gland minus CTV_40 (CTV_25) will be prescribed to 5 Gy x 5 fractions at the 95% isodose line.
Drug: Androgen Deprivation Therapy (ADT) — ADT would be given 0-1 months prior to planned SBRT to the prostate for total of 4-6 months. ADT will be administered via Leuprolide or Degarelix monthly injections or daily Relugolix pills.

SUMMARY:
The purpose of this study is to assess the impact of prostate-specific membrane antigen/positron emission tomography (PSMA/PET)-informed magnetic resonance (MR)-guided radiation therapy on serious toxicity outcomes in patients with biopsy-proven locally radiorecurrent prostate cancer. The primary aim is to evaluate the safety of delivering MR-Linac-guided stereotactic body radiotherapy (SBRT) after prior prostate external beam radiotherapy for recurrent disease, and assess urinary toxicity outcomes at 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older male participants
2. Biopsy proven intraprostatic prostate cancer after prior definitive external beam radiotherapy (moderate hypofractionation or Stereotactic Body Radiation Therapy (SBRT) acceptable).

   a. NOTE: Seminal vesicle involvement allowed
3. Pathology confirming recurrent disease must have evidence of viable cancer as indicated with pathology interpretation where a Gleason score can be assigned
4. Serum testosterone ≥ 50 ng/dL determined within 2 months prior to enrollment

   a. Prior Androgen Deprivation Therapy (ADT) use acceptable if testosterone level >50ng/dL
5. At least 4 weeks must have elapsed from major surgery
6. Karnofsky Performance Scale (KPS) ≥ 80% or Eastern Cooperative Oncology Group (ECOG) 0-1
7. Prostate size as determined on MRI to be < 90 cc.
8. International Prostatism Symptom Score (IPSS) ≤ 20
9. Patient must be available for follow-up. After 2 years of follow-up, upon completion of post-treatment biopsy, telephone, and chart review-based follow-up will be acceptable for up to 5 years
10. Presence of a T2 and/or DWI-visible prostatic lesion on mpMRI

    a. NOTE: Lesion visible on MRI required for enrollment but PSMA/PET avid lesion not required
11. Satisfy all MRI screening criteria and be willing to fill out the standard MRI screening form

Exclusion Criteria:

1. History of prostate brachytherapy (low dose rate or high dose rate)
2. Actively undergoing androgen deprivation therapy and/or anti-androgens at time of enrollment
3. CT or MRI or PET scan evidence of extraprostatic disease
4. Patients with one or more positive lymph nodes considered suspicious as determined by clinical assessment on MRI or CT or PET scan
5. History of another malignancy within the previous 2 years except for the following: adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, currently in complete remission, or any other cancer that has been in complete remission for at least 3 years
6. Patients with Crohn's disease or ulcerative colitis
7. MRI ineligibility due to: the presence of a cardiac pacemaker, defibrillator, or other implanted metallic or electronic device which is considered MR unsafe; severe claustrophobia; inability to lie flat for the duration of the study; etc.
8. Metallic implant or device in the pelvis that might distort the local magnetic field and compromise quality of mp-MRI
9. Lateral pelvic separation greater than 50 cm and/or anterior-posterior separation greater than 35 cm which are incompatible with MRCAT reconstruction
10. Contra-indications to receiving gadolinium contrast or PSMA radioligand
11. Karnofsky Performance Scale (KPS) < 80 or ECOG 2+
12. Grade 3 or higher toxicity experienced after the initial course of External Beam Radiation Therapy (EBRT)
13. Disease free interval < 2 years
14. Hx of Transurethral Resection Of Prostate (TURP) within the year
15. Prior high-intensity focused ultrasound (HIFU) or Cryotherapy
16. Prior history of urethral stricture
17. Unable to give informed consent
18. Unable to complete quality of life questionnaires

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2029-08-02 (Estimated)

PRIMARY OUTCOMES:
Late toxicity (after 90 days) radiation-associated genitourinary (GU) and gastrointestinal (GI) events | Month 24
  A serious toxicity event will be defined as any Grade 3 or higher genitourinary or gastrointestinal toxicity, based on NCI CTCAE v5.0.

SECONDARY OUTCOMES:
Acute toxicity (occurring within 90 days of the treatment) radiation-associated genitourinary (GU) and gastrointestinal (GI) events | Month 24
  A serious toxicity event will be defined as any Grade 3 or higher genitourinary or gastrointestinal toxicity, based on NCI CTCAE v5.0.
Biochemical progression free survival | Month 24
  From the time after treatment until the prostate-specific antigen (PSA) level rises, indicating a potential return of cancer.
Distant metastasis-free survival (DMFS) | Month 24
  Distant metastasis-free survival (DMFS) the time from end of treatment until the first instance of distant metastasis or death, whichever occurs first.
Radiographic treatment response rate of target intra-prostatic lesion | Month 24
  Radiographic treatment response rate is the patients whose tumors show a reduction in size or other measurable changes on imaging scans after receiving treatment.
Expanded Prostate cancer Index Composite (EPIC-26) Short Form score | Month 24
  The EPIC-26 short form scores range from 0 to 100 for each of its five domains (urinary incontinence, urinary irritative/obstructive, bowel, sexual, and hormonal). Higher scores indicate better health-related quality of life (HRQOL) within that domain.
International prostate symptom score index (IPSS) score | Month 24
  The IPSS index is a seven-item questionnaire designed to assess urinary functioning, specifically urinary frequency, nocturia, weak urinary stream, hesitancy, intermittence, incomplete emptying, and urgency. Questions are rated on a six-point Likert scale, scores range from 0 to 35, with higher scores indicating more severe urinary symptoms. Scores are categorized as mild (0-7), moderate (8-19), or severe (20-35).
International Index of Erectile Function (IIEF) score | Month 24
  The IIEF 5 form is a 5-item questionnaire used to assess erectile function and diagnose erectile dysfunction (ED). Participant rate their responses using a 6-point Likert Scale (0-5). Scores range from 5 to 25. Scores are categorized as follows: 5-7 (severe ED), 8-11 (moderate ED), 12-16 (mild to moderate ED), 17-21 (mild ED), and 22-25 (no ED)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zelefsky, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: Michael.zelefsky@nyulangone. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Michael.zelefsky@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.